CLINICAL TRIAL: NCT04247555
Title: Cervix Monitor for Elasticity and Length Measurements
Brief Title: Cervix Monitor for Detection Conditions Leading to Spontaneous Preterm Delivery
Acronym: CM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Advanced Tactile Imaging, Inc. (Industry)
Collaborators: Rutgers, The State University of New Jersey (Other); St. Luke's Hospital and Health Network, Pennsylvania (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: CM02; R44HD090793 (NIH)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

SUMMARY:
Preterm birth is a leading cause of neonatal mortality despite of numerous advances and intensive research in perinatal medicine. Almost one million children die every year due to the complications of preterm birth and rates are on the rise. Of the 14 million survivors per year, most face a lifetime of disability, including learning disabilities, visual and hearing impairments. The majority of preterm birth happen spontaneously (SPTD) which is often a multi factorial event, precocious cervical softening, shortening and dilatation are a common underlying factor. In the scope of this project the investigators propose to develop and clinically validate a new device, Cervix Monitor (CM), for detecting cervix conditions leading to SPTD and its risk assessment.

DETAILED DESCRIPTION:
SPTD is closely related to a premature cervical ripening. The scientific basis for the proposed project is that the elasticity modulus of a cervix is a more sensitive parameter characterizing the stage of cervical ripening. The main component of the cervical tissue is collagen. Cervical ripening is the result of realignment of collagen, degradation of collagen cross-linking due to proteolytic enzymes. These processes affect the elasticity modulus of the cervical tissue. Therefore, assessment of cervix by a device (CM) measuring cervical elasticity (stiffness) and cervical length (effacement) appears to be an adequate approach for identifying pregnant women at high risk of SPTD. The CM is based on measuring applied pressure to the cervix by a tactile sensor array (stress data) and ultrasound measurement of cervix length (strain data). Tactile and ultrasound sensors are allocated on the tip of the measuring part of vaginal probe. The discovery of novel bio markers that could reliably identify women who will subsequently deliver preterm, may allow for timely medical intervention and targeted therapeutic treatments aimed at improving maternal and fetal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age from 24 to 28 weeks at time of Cervix Monitor measurement
* Singleton in the current pregnancy

Exclusion Criteria:

* Fatal anomaly
* History of fetal reduction in the current pregnancy to the singleton gestation
* Preterm rapture of membranes
* Current or planned cervical cerclage
* Planned indicated preterm delivery
* Active known cancer of the colon, rectum wall, cervix, vaginal, uterus or bladder
* Ischemic heart disease and or arrhythmia
* Active skin infection or ulceration within the vaginal/vulva (Herpes infection)

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women with gestational age from 24 to 28 weeks.
Study Population: Woman at 24 to 28 weeks of pregnancy scheduled for a regular examination at the Divisions of Maternal Fetal Medicine will be considered eligible for this study enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Cervix elasticity | During examination procedure
  Units measurement of elasticity in kPa
Cervix Length | During examination procedure
  Units of measurement of length in mm

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Egorov, PhD, Principal Investigator — Advanced Tactile Imaging, Inc.
Locations (2):
- United States (2):
  - Rutgers The State University Of New Jersey, New Brunswick, New Jersey
  - St. Luke's University Health Network Department of Obstetrics and Gynecology, Division of Maternal Fetal Medicine (MFM), Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egorov V, Rosen T, van Raalte H, Kurtenoks V. Cervical Characterization with Tactile-Ultrasound Probe. Open J Obstet Gynecol. 2020 Jan;10(1):85-99. doi: 10.4236/ojog.2020.101008. Epub 2020 Jan 8. PMID 32133244
- [Background] Lucente V, van Raalte H, Murphy M, Egorov V. Biomechanical paradigm and interpretation of female pelvic floor conditions before a treatment. Int J Womens Health. 2017 Aug 3;9:521-550. doi: 10.2147/IJWH.S136989. eCollection 2017. PMID 28831274